CLINICAL TRIAL: NCT00357539
Title: Comparison of the Ocular Tolerance, the Safety and the Ocular Pharmacokinetics After One Drop of Three Different Concentrations of T1225 (0.5% - 1.0% - 1.5%) in 48 Healthy Volunteers
Brief Title: Safety and Ocular Pharmacokinetics After 1 Drop of T1225 0.5, 1 and 1.5% in 48 Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1225-PI1-09/01(F)
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: Eye Infections, Bacterial
MeSH Terms: conditions — Eye Infections, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin (T1225)

SUMMARY:
To compare the ocular tolerance, safety and ocular pharmacokinetics of 3 concentrations (0.5% - 1.0% - 1.5%) and the vehicle of T1225.

DETAILED DESCRIPTION:
The present phase I clinical trial was performed in order to investigate the ocular tolerance, safety and the ocular pharmacokinetics of a single administration of T1225 eye drops (0.5%, 1.0%, or 1.5%) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 45 years old;
* Written informed consent;
* Healthy volunteers (without any ocular symptom);
* Normal ocular examination in both eyes (corrected visual acuity (VA) >= 6/10 - slit lamp examination without clinical relevant abnormalities - tear break-up time (BUT) >= 10 seconds - lachrymal secretion in the Schirmer test >= 10 mm in 5 minutes - lissamine green test total score < 4).

Exclusion Criteria:

* Ocular trauma, infection or inflammation within the last 3 months;
* Conjunctival hyperaemia score >= 2, watering score >= 2, folliculo-papillary conjunctivitis score >= 2, number of fluorescein-stained punctuations >= 10;
* Blepharitis, conjunctivitis, uveitis;
* Ocular laser treatment within the last 3 months;
* Ocular surgery, including LASIK and PRK, within the last 12 months;
* Topical ocular treatment during the last month;
* Ocular antibiotics within the last 7 days;
* Medication during the study (except paracetamol and contraceptives).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2002-02; Study Completion 2002-03

PRIMARY OUTCOMES:
Subjective ocular symptoms
Objective ocular symptoms

SECONDARY OUTCOMES:
Systemic adverse events
Ocular adverse events
Ocular pharmacokinetic

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Professor, Principal Investigator — Unité de Pharmacologie Clinique - Clermont-Ferrand (France)
Locations (1):
- Unité de Pharmacologie Clinique, Clermont-Ferrand, France